CLINICAL TRIAL: NCT01904305
Title: Clinician Ability to Predict the Presence of Nosocomial Pneumonia Based on Macroscopic Examination of Bronchoscopic Findings in Critically Ill Surgical Patients
Brief Title: Clinician Ability to Predict the Presence of Nosocomial Pneumonia Based on Bronchoscopic Findings
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Bryce Robinson, MD, Assistant Clinical Professor, University of Cincinnati
Other Study IDs: Robinson-2010-01
Record Dates: First submitted 2011-11-18; First posted 2013-07-22 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Pneumonia
Keywords: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Standard lavage specimens collected as part of standard of care and submitted for laboratory evaluation
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients receiving bronchoscopy: Patients suspected of having pneumonia received bronchoscopy to examine the lungs and to capture alveolar lavage culture

SUMMARY:
This study aims to determine whether interpretations of bronchoscopic results enable physicians to successfully predict the presence of pneumonia in traumatically injured patients.

DETAILED DESCRIPTION:
This study aims to determine whether interpretations of bronchoscopic results enable physicians to successfully predict the presence of pneumonia in traumatically injured patients. Bronchoscopies will be videotaped. The clinician doing the procedure will make prediction as to whether the patient, in fact, has pneumonia. In addition, at least one other physician will view the videotape and predict whether the patient has pneumonia.

Once laboratory results are available, the physician predictions will be compared against the definitive laboratory determination

ELIGIBILITY:
Inclusion Criteria:

* Critical Care staff and fellows of the Departments of Anesthesia and Surgery

Exclusion Criteria:

* Refusal of consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physicians working in the Surgical Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Presence or absence of hospital-acquired pneumonia | At first clinical suspicion of pneumonia. Average of hospital Day 4
  When pneumonia is suspected, patient with undergo bronchoscopy. BAL specimens will be submitted to laboratory testing. Laboratory results are the definitive indication of pneumonia, or lack thereof.

CONTACTS AND LOCATIONS:
Overall Officials: Bryce RH Robinson, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University Hospital, Cincinnati, Ohio, United States